CLINICAL TRIAL: NCT03047161
Title: Electrophysiology of Fetal Arrhythmia
Acronym: fMCG
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2013-0362 Stage 3; A534800 (Other: UW Madison); SMPH\MEDICAL PHYSICS (Other: UW Madison); 2R01HL063174-19A1 (NIH); Protocol Version 7/16/2024 (Other: UW Madison); R44HL160257 (NIH)
Record Dates: First submitted 2017-02-02; First posted 2017-02-08 (Estimated); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Fetal Arrhythmia
Keywords: magnetocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — fetal magnetocardiography and fetal echocardiography recordings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- High-risk pregnancy: abnormal fetal heart rate or rhythm or risk of abnormal fetal heart rate or rhythm
  Interventions: Device: fetal MCG
- Uncomplicated pregnancy: uncomplicated pregnancy
  Interventions: Device: fetal MCG

INTERVENTIONS:
Device: fetal MCG — assess fetal heart rate and rhythm

SUMMARY:
Fetal research and clinical practice has been hampered by a lack of suitable investigational techniques. Currently, ultrasound is the only widely used method of studying fetal anatomy and physiology, but it has significant limitations for assessment of cardiac rhythm. The proposed study will allow the investigators to evaluate fetal magnetocardiography (fMCG) as a new tool for the study of normal and abnormal fetal heart rate and rhythm.

DETAILED DESCRIPTION:
Purpose

Fetal research and clinical practice has been hampered by a lack of suitable investigational techniques. Currently, ultrasound is the only widely used method of studying fetal anatomy and physiology, but it has significant limitations for assessment of cardiac rhythm. The purpose of the proposed study is to utilize fMCG, the magnetic analog of fetal ECG, to characterize the heart rate and rhythm patterns of fetuses with fetal arrhythmia or at risk of fetal arrhythmia. The study is not intended to be a pivotal study. The subject device is already cleared for clinical use for recording of fetal rhythm; however, FDA has determined that an IDE is required for the proposed study. The study is expected to last approximately 6 years

The Tristan 624 is housed within the magnetically shielded room in the Biomagnetism Laboratory located within the Wisconsin Institutes for Medical Research on the University of Wisconsin-Madison campus.

Protocol

Facilities

The UW Biomagnetism Lab is located within the Wisconsin Institutes for Medical Research, a state-of-the-art translational research facility adjacent to UW Hospitals and Clinics. The study sponsor, Ronald Wakai, PhD, Professor of Medical Physics, is the Laboratory Director. Within the laboratory, medical supervision is provided by Janette Strasburger, MD. The facility is directly adjacent to UW Hospital. An emergency response plan is in place for the facility and for the Biomagnetism Lab. In the study of over 700 pregnancies thus far, the emergency response plan has not been needed.

Subject cohort

The investigators plan to study a total of 300 subjects: 75 will be pregnant women with uncomplicated pregnancies and 225 will be pregnant women with pregnancies complicated by fetal arrhythmia or a condition that puts the fetus at risk of fetal arrhythmia. These cases are considered "high-risk" due to the presence of or risk of serious arrhythmia to the fetus. It will take approximately 5 years from the start of data collection to recruit the subjects and collect and analyze the data. The pregnant mothers will be age 18 or older. They will be studied as early as 15 weeks' gestation and may be asked to return about once every 4 weeks, if their physician determines that additional fMCG studies are necessary.

Inclusion criteria for normal subjects. The pregnant women subjects must be at least 12 weeks pregnant and at least 18 years old. They must have uncomplicated pregnancies.

Exclusion criteria for normal subjects. The pregnant women subjects will be excluded if they are earlier than 12 weeks pregnant or younger than age 18. The 510(k) summary lists no exclusions for the use of the subject device.

Inclusion criteria for high-risk subjects. The pregnant women subjects must be at least 15 weeks pregnant and at least 18 years old. The primary inclusion criterion is diagnosis of serious fetal arrhythmia, which is defined as sustained low or high heart rate. Low heart rate, or bradycardia, and high heart rate, or tachycardia, are based on normative values for gestation (usually below 110 -120 beats/min, or above 160-180 beats/min). Intermittent bradycardia or tachycardia and frequent and/or complex ectopy (irregular rhythm) are also important to detect because these arrhythmias may become incessant over the course of pregnancy and have implications for patient management. Abnormal repolarization, such as long QT syndrome (LQTS), is another important class of arrhythmia. Fetuses with a family history of LQTS or a suspicious rhythm (low heart rate, intermittent AV block, or ventricular tachycardia) will also be studied.

Exclusion criteria for high-risk subjects. The pregnant women subjects will be excluded if they are earlier than 15 weeks pregnant or younger than age 18. High-risk subjects cannot participate if their physician does not grant permission for them to participate in the study. Again, the 510(k) summary lists no exclusions for the use of the subject device.

Recruitment methods

* Women age 18 or older with uncomplicated pregnancies will be recruited by placing posters in local perinatal clinics. When prospective subjects call, the study is described to them and they are asked if they have any high-risk conditions that might affect their participation. If any issues arise, Dr. Wakai in consultation with Dr. Strasburger determines whether they are appropriate to study. Informed consent will be obtained at the time of study by Dr. Wakai or one of his associates. Normal subjects will be invited to return for follow up sessions up to 5 times.
* Pregnancies complicated by fetal arrhythmia and or at risk of fetal arrhythmia will be recruited by Dr. Janette Strasburger, Medical College of Wisconsin. She will screen the subjects, explain the procedure, counsel them, and recruit them for the study prior to referring them on to Dr. Wakai. These patients are already being clinically evaluated and it is not anticipated that advertising for participants or posting of flyers will be required. In addition to patients from Madison, Milwaukee and Chicago, high-risk patients from across the country may be enrolled in the study. In these cases the patient's physician has contacted the investigators because he/she believes fMCG may be beneficial for clinical care. These high-risk subjects are screened for appropriateness by Dr. Strasburger, who will consult with the patient's physician in order to determine whether the risk of travel to Madison is reasonable. Informed consent will be obtained at the time of study at the Biomagnetism Lab by Dr. Wakai or one of his associates.
* There are no inclusion or exclusion criteria based on race or ethnicity. Informed Consent
* Informed consent requirements and regulations relating to informed consent will be followed. Informed consent will be obtained prior to performing any study-related activities.
* Prior to signing a consent form, subjects are given a tour of the lab, the experimental procedures are described to them, and their questions are answered. For all subjects, consent and HIPAA authorization will be obtained by the PI or one of his representatives at the time of study.

Subject preparation

The subject is asked to remove all metal and magnetic objects (e.g. watches, glasses, jewelry, coins) from her person and change into a patient gown. The subject lies on a patient table in a magnetically shielded room throughout the study. An intercom system allows verbal communication at all times and the subject can be observed through an aperture in the room.

Data Acquisition

Ultrasound. An ultrasound exam will be performed by Dr. Strasburger to assess the heart rhythm of the fetus. The exam will be performed according American Society of Echocardiography (ASE) standards for fetal arrhythmia.

fMCG recording. The SQUID detector is placed over the maternal abdomen near the location of the fetal heart. Several 10-minute recordings are made, repositioning the detector between recordings,

Data analysis.

fMCG

After the recordings are digitally filtered to band-limit the signal, signal processing techniques are applied to remove maternal interference. Maternal heart rate is evaluated. The fetal QRS complexes are detected using autocorrelation. Fetal heart rate tracings are calculated from the RR intervals, and actogram tracings are derived from the instantaneous amplitude of the QRS complex, which changes in response to fetal trunk movement. Averaged fMCG waveforms are computed to increase the signal-to-noise ratio. The data are organized into a report. The reports consist of 1) fetal heart rate and actogram tracings, 2) averaged fMCG waveforms, and 3) fMCG rhythm strips. Rhythm interpretation and clinical diagnosis is based on assessment of these data. The fetal heart rate tracings are used to identify periods of abnormal heart rate, corresponding to bradycardia, tachycardia, or ectopy. The fetal heart rate tracings and actograms can be used to assess heart rate reactivity, which is an association between fetal heart rate acceleration and fetal movement. The fetal heart rate tracings can also be used to assess fetal heart rate variability with high precision.

The averaged waveforms are used to measure waveform intervals-PR, QRS, QTc-which can be used to detect abnormalities in AV conduction, ventricular conduction, and repolarization. The intervals are defined the same way as for the ECG: PR interval is measured from the onset of the P-wave to the onset of the QRS complex; QRS interval measures the duration of the QRS complex; QT interval is measured from the onset of the QRS complex to the termination of the T-wave; and the corrected QT interval, QTc, corrects the QT interval for heart rate by dividing by the square root of the RR interval, measured in seconds. The intervals are compared with historical norms. The rhythm strips are used to diagnose rhythm abnormalities in a similar way as an ECG, based on the timing and morphology of the waveform components.

For fetal arrhythmia and other high-risk subjects, the results will be interpreted by Dr. Strasburger, who sends the report to and discusses the results with the referring physician. In order to protect the confidentiality of the subject, the data will be sent in electronic files labeled with an identification number, but the referring physician and Drs. Strasburger will be made aware of the identity of the subject (patient).

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated pregnancy at gestational age >12 weeks
* pregnancy complicated by abnormal fetal heart rate or rhythm or risk of abnormal fetal heart rate or rhythm at gestational age >15 weeks

Exclusion Criteria:

* uncomplicated pregnancy <12 weeks gestation
* pregnancy complicated by abnormal fetal heart rate or rhythm or risk of abnormal fetal heart rate or rhythm at gestational age <15 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Uncomplicated pregnancies and pregnancies complicated by abnormal fetal heart rate or rhythm or risk of abnormal fetal heart rate or rhythm
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2017-02-07 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Rhythm assessment | after 15 weeks gestation
  fetal MCG rhythm assessment

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Wakai, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wacker-Gussmann A, Tardelli G, Cuneo BF, Strasburger JF, Wakai RT. Fetal Conduction Disease and Arrhythmia in Ebstein's Anomaly and Tricuspid Valve Dysplasia Assessed by Fetal Magnetocardiography. J Am Heart Assoc. 2025 Aug 5;14(15):e043614. doi: 10.1161/JAHA.125.043614. Epub 2025 Jul 29. PMID 40728160
- [Derived] Strand S, Strasburger JF, Cuneo BF, Wakai RT. Complex and Novel Arrhythmias Precede Stillbirth in Fetuses With De Novo Long QT Syndrome. Circ Arrhythm Electrophysiol. 2020 May;13(5):e008082. doi: 10.1161/CIRCEP.119.008082. Epub 2020 May 18. PMID 32421437